CLINICAL TRIAL: NCT02622828
Title: Increasing the Winter Community Participation of Older Adult Wheelchair Users
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Unable to recruit needed participants
Sponsor: University of Manitoba (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: H2015:132
Record Dates: First submitted 2015-12-01; First posted 2015-12-07 (Estimated); Results first posted 2019-10-04 (Actual); Last update posted 2019-10-04 (Actual); Status verified 2016-08

CONDITIONS: Frail Elderly
Keywords: wheelchairs; social participation

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Behavioural (Other): Participant-identified community based activity
  Interventions: Behavioral: Participant-identified community based activity

INTERVENTIONS:
Behavioral: Participant-identified community based activity — The Canadian Occupational Performance Measure (COPM) is a client-centered outcome measure designed to detect changes in performance and satisfaction in occupations that the individual has self-identified as being important and difficult to perform. The COPM will be used to set self-identified, community-based activities as treatment goals.

SUMMARY:
The purpose of this study is to examine whether intervention strategies targeted at the level of the environment (e.g. improving access to community based leisure groups, transportation) can successfully promote the community participation experiences of community-dwelling older adult Manitobans who use wheelchairs in the winter.

DETAILED DESCRIPTION:
There is strong evidence to support that community-dwelling older adults who are able to maintain their involvement in social, recreational, spiritual and physical activities experience positive effects on their health and quality of life. While winter creates challenges to community participation for many Manitobans, these difficulties are magnified for older adults and particularly for older adults who use wheelchairs. The aim of this study is to explore ways to improve or maintain community participation of community-dwelling older adults who use wheelchairs in the winter. Using a single-subject design, five older adult Manitobans who are wheelchair users will each select three community-based participation goals to work on throughout the winter months. Each older adult participant will work with an occupational therapist to receive individually-focused interventions aimed at increasing his or her community participation. The investigators will use a client-centered outcome measure designed to detect changes in performance and satisfaction in the goals that the individual has self-identified as being important to him or her, yet difficult to perform. The findings of this study will help determine the feasibility of conducting a larger scale study that would include a greater number of older adult Manitobans. Older adult wheelchair users in Manitoba bear a disproportionate burden in the winter when aging, mobility limitations, and weather coincide to create conditions that make community participation exceedingly difficult. It is important to the health and well-being of older adult Manitobans to find effective ways to promote community engagement throughout the winter months.

ELIGIBILITY:
Inclusion Criteria:

* Age 70 or older, user of a manual or power wheelchair or scooter for outdoor mobility
* Self-identifies a reduction in community participation throughout the winter months
* Community-dwelling
* Lives within the perimeter of Winnipeg.

Exclusion Criteria:

* Geriatric Depression Scale-SF score of 6 or more
* Montreal Cognitive Assessment score of 25 or less

Min Age: 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Older Adult
Enrollment: 4 (Actual)
Dates: Start 2015-12-01 (Actual); Primary Completion 2017-09-15 (Actual); Study Completion 2017-09-15 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jacquie Ripat, PhD, Principal Investigator — University of Manitoba
Locations (1):
- University of Manitoba, Winnipeg, Manitoba, Canada

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Behavioural
Started | 4
Completed | 1
Not Completed | 3
Not completed — participant withdrew | 3

BASELINE CHARACTERISTICS:
Arm/Group | Behavioural
Number analyzed (Participants) | 4
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 0
  >=65 years | 4
Age, Continuous [Median (Full Range); unit: years] — Population: participants enrolled but did not complete study
  years | 75 [70 to 80]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3
  Male | 1
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0
  Not Hispanic or Latino | 0
  Unknown or Not Reported | 4
Region of Enrollment [Number; unit: participants]
  Canada | 4
Canadian Occupational Performance Measure [Number; unit: units on a scale] — The Canadian Occupational Performance Measure (COPM) is a client-centered outcome measure designed to detect changes in performance and satisfaction in occupations that the individual has self-identified as being important and difficult to perform. At baseline, participants self-identify 5 occupation (activity-based) goals and rate performance and satisfaction on each on a likert scale from 1 (low performance/satisfaction) to 10 (high performance/satisfaction). A performance and satisfaction sub-score are calculated for each person based on the mean score of the 5 items. Population: Data not collected for this assessment

OUTCOME MEASURES:

1. Primary Outcome: Change in Occupational Performance Using the The Canadian Occupational Performance Measure (COPM) at 5 Months
Description: The Canadian Occupational Performance Measure (COPM) is a client-centered outcome measure designed to detect changes in performance and satisfaction in occupations that the individual has self-identified as being important and difficult to perform. The COPM has well-established psychometric properties and will be used as the primary outcome measure and will be used to set treatment goals, determine baseline stability, and detect change in performance of, and satisfaction with, the goals.
Time Frame: Initial and 5 month follow up
Population: data were not collected
Arm/Group | Behavioural
Number analyzed (Participants) | 0

2. Secondary Outcome: World Health Organization Disability Assessment Schedule 2.0 (WHO-DAS2)
Description: The WHO-DAS 2.0 is a generic self-report health status measure, linked to the concepts of health and disability outlined in the International Classification of Functioning, Disability and Health and is intended to identify limitations in six domains with 36 items, including self-care, and community and social functioning experienced over the past 30 days. The WHO-DAS 2.0 is responsive to change, has excellent internal consistency, established content validity, and high convergent validity. The WHO-DAS 2.0 will be used to identify changes in overall health status that occur through the study. Uses a scale of 1-5 - 1=no difficulty and 5=extreme difficulty or cannot do. Sum of items within each domain are then summed across the 6 domains to result in a general disability summary score, converted to a metric from 0-100 with higher score indicating more disability.
Time Frame: Initial and 5 month follow-up
Population: data were not collected
Arm/Group | Behavioural
Number analyzed (Participants) | 0

ADVERSE EVENTS:
Time Frame: 2 years
Arm/Group | Behavioural
All-Cause Mortality (participants affected / at risk) | 0/4
Serious Adverse Events (participants affected / at risk) | 0/4
Other Adverse Events (participants affected / at risk) | 0/4

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2015-10-02): https://cdn.clinicaltrials.gov/large-docs/28/NCT02622828/Prot_SAP_000.pdf